CLINICAL TRIAL: NCT06456268
Title: Clinical Evaluation of an External Neuromodulation Device (VibraCool) to Reduce Pain and Opioid Use After Anterior Cruciate Ligament Reconstruction (ACLR)
Brief Title: VibraCool Device to Reduce Pain and Opioid Use After Anterior Cruciate Ligament Reconstruction (ACLR)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Lauren H. Redler, Assistant Professor of Orthopedic Surgery, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAAU3696
Record Dates: First submitted 2024-06-08; First posted 2024-06-13 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: ACL; Opioid Use; Cryotherapy Effect; Vibration; Exposure; Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinded data will be provided to the statistician w/o reference to specific treatment arms
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Standard Ice packs (Active Comparator): Standard ice packs applied to knee for 20 minutes a day three times a day
  Interventions: Device: Standard ice packs
- Cryocompression device (Active Comparator): Cryocompression device (Game Ready, Bregs) with ice placed into the device and applied to knee for 20 minutes a day, three times a day
  Interventions: Device: Cryocompression (Game Ready, Bregs) device
- VibraCool (Experimental): FDA-approved VibraCool mechanical stimulation and neuromodulatory therapeutic device with ice placed into it and applied to knee for 20 minutes a day, three times a day
  Interventions: Device: VibraCool mechanical stimulation and neuromodulatory therapeutic device

INTERVENTIONS:
Device: VibraCool mechanical stimulation and neuromodulatory therapeutic device — Multiple studies have shown that vibration sources applied to muscles prior to exercise reduced soreness and lactate dehydrogenase production, and increased range of motion at 48 and 72 hours. Acute pain results from fast A nerves transmitting nociceptive information to the dorsal column, where the substantia gelatinosa's interneurons prioritize competing A mechanoreceptor and C-fibers to slow pain transmission. One study observed that stimulation of A mechanoreceptors "shut the gate" on pain transmission, an inhibitory mechanism known as "gate control". Multiple physical methodologies leverage gate control physiology for pain relief, such as vibratory massage therapy and electrical stimulation to varying degrees. However, the use of vibratory massage to improve pain control and reduce opioid use following ACLR has not been well studied, and to our knowledge there are no randomized control trials (RCTs) evaluating the use of this modality compared to standard ice or cryocompression.
  Arms: VibraCool
Device: Cryocompression (Game Ready, Bregs) device — Cryotherapy has also been used as an adjunctive post-operative therapy to reduce pain and inflammation following anterior cruciate ligament reconstruction (ACLR). It has been shown to decrease local metabolism, resulting in reduced pain and inflammation. Multiple studies have shown the benefits of using cryotherapy after ACLR, and more recently dynamic intermittent compression has been shown to improve circulation while reducing the risk of skin necrosis associated with static permanent compression. A recent meta-analysis including ten RCTs found significant reductions in post-operative VAS pain scores and breakthrough opioid consumption when using cryotherapy, such as Game Ready or Breggs ice therapy, following ACLR.
  Arms: Cryocompression device
Device: Standard ice packs — Cold also provides peripheral gate-control relief via small, slow C-Fibers that transmit low level pain. In addition to local pain relief, intense cold can raise the A pain threshold distant to the location. The mechanism has been called descending or diffuse noxious inhibitory relief, or more recently conditioned pain modulation (CPM). Injections, aches, and infiltration of local anesthesia and dermal fillers are relieved by applying cold. For acute injury, near freezing cold relieves pain by suppressing the local metabolic production of inflammation and concomitant tissue ischemia from hypoxia due to the increased metabolic rate.
  Arms: Standard Ice packs

SUMMARY:
The goal of this project is to test the effects of the VibraCool mechanical stimulation neuromodulatory therapeutic device on post-operative pain and opioid use following anterior crucitate ligament reconstruction (ACLR), and thus residual opioids in circulation.

ELIGIBILITY:
Inclusion Criteria:

* Underwent ACL reconstruction

Exclusion Criteria:

* Pediatric iliotibial band ACL reconstruction (known to cause significantly more pain)
* Non-english speakers (limitations of our study group)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Score (VAS) for pain | First 7 post-operative days
  Scale of 0 to 10, with 10 being the worst pain and 0 being no pain. Will record daily mean VAS pain scores over the first seven post-operative days
Opioid use | First 3 post-operative days
  Percent of patients discontinuing opioid use by or on post-operative day three, compared to those who continue after day three

SECONDARY OUTCOMES:
Mean reduction in opioid use in mg of morphine equivalents per day | First 7 post-operative days
  mean reduction in opioid use in milligrams of morphine equivalents per day (MMOD) of 30% from patients not using the device over the 7-day period
Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference score | First 7 post-operative days
  PROMIS is a computerized adaptive patient-reported test to measure interference of pain in everyday functioning. The raw score is converted to a T-score metric in which 50 is the mean and 10 is the standard deviation. Higher T-scores represent increased pain interference.

CONTACTS AND LOCATIONS:
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
None will be shared

REFERENCES:
- [Background] Bartels K, Mayes LM, Dingmann C, Bullard KJ, Hopfer CJ, Binswanger IA. Opioid Use and Storage Patterns by Patients after Hospital Discharge following Surgery. PLoS One. 2016 Jan 29;11(1):e0147972. doi: 10.1371/journal.pone.0147972. eCollection 2016. PMID 26824844
- [Background] Webster BS, Verma SK, Gatchel RJ. Relationship between early opioid prescribing for acute occupational low back pain and disability duration, medical costs, subsequent surgery and late opioid use. Spine (Phila Pa 1976). 2007 Sep 1;32(19):2127-32. doi: 10.1097/BRS.0b013e318145a731. PMID 17762815
- [Background] Bleakley C, McDonough S, MacAuley D. The use of ice in the treatment of acute soft-tissue injury: a systematic review of randomized controlled trials. Am J Sports Med. 2004 Jan-Feb;32(1):251-61. doi: 10.1177/0363546503260757. PMID 14754753
- [Background] Clarke H, Soneji N, Ko DT, Yun L, Wijeysundera DN. Rates and risk factors for prolonged opioid use after major surgery: population based cohort study. BMJ. 2014 Feb 11;348:g1251. doi: 10.1136/bmj.g1251. PMID 24519537
- [Background] Crystal NJ, Townson DH, Cook SB, LaRoche DP. Effect of cryotherapy on muscle recovery and inflammation following a bout of damaging exercise. Eur J Appl Physiol. 2013 Oct;113(10):2577-86. doi: 10.1007/s00421-013-2693-9. Epub 2013 Jul 20. PMID 23873339
- [Background] Davey MS, Hurley ET, Anil U, Moses A, Thompson K, Alaia M, Strauss EJ, Campbell KA. Pain Management Strategies After Anterior Cruciate Ligament Reconstruction: A Systematic Review With Network Meta-analysis. Arthroscopy. 2021 Apr;37(4):1290-1300.e6. doi: 10.1016/j.arthro.2021.01.023. Epub 2021 Jan 28. PMID 33515736
- [Background] Scully RE, Schoenfeld AJ, Jiang W, Lipsitz S, Chaudhary MA, Learn PA, Koehlmoos T, Haider AH, Nguyen LL. Defining Optimal Length of Opioid Pain Medication Prescription After Common Surgical Procedures. JAMA Surg. 2018 Jan 1;153(1):37-43. doi: 10.1001/jamasurg.2017.3132. PMID 28973092
- [Background] Hollins M, Roy EA, Crane SA. Vibratory antinociception: effects of vibration amplitude and frequency. J Pain. 2003 Sep;4(7):381-91. doi: 10.1016/s1526-5900(03)00714-4. PMID 14622680
- [Background] Khanna A, Gougoulias N, Maffulli N. Intermittent pneumatic compression in fracture and soft-tissue injuries healing. Br Med Bull. 2008;88(1):147-56. doi: 10.1093/bmb/ldn024. Epub 2008 Jul 1. PMID 18596049
- [Background] Benedetti MG, Boccia G, Cavazzuti L, Magnani E, Mariani E, Rainoldi A, Casale R. Localized muscle vibration reverses quadriceps muscle hypotrophy and improves physical function: a clinical and electrophysiological study. Int J Rehabil Res. 2017 Dec;40(4):339-346. doi: 10.1097/MRR.0000000000000242. PMID 28723717

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-14): https://cdn.clinicaltrials.gov/large-docs/68/NCT06456268/Prot_SAP_000.pdf